CLINICAL TRIAL: NCT05025306
Title: Healing Effect of Ziziphus Honey on Extracted Tooth Socket in Humans by Evaluating the Levels of BMP-2 and OPN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Postgraduate Medical Institute, Lahore (Other)
Responsible Party: Principal Investigator, Momina khalid, Principal investigator, Postgraduate Medical Institute, Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PGMILahore
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Healing Wound
MeSH Terms: interventions — Honey

STUDY DESIGN:
Intervention Model Description: randomized controlled trial with simple random sampling technique
Who Masked: Participant
Masking Description: Participants were not aware of the intervention used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): only atraumatic extractions were done, honey was not applied
- experimental group (Experimental): ziziphus honey was applied into the sockets after tooth extractions in experimental group
  Interventions: Drug: ziziphus honey

INTERVENTIONS:
Drug: ziziphus honey — ziziphus honey obtained form ziziphus spina-christi trees also called sidr tree
  Other Names: sidr honey; honey
  Arms: experimental group

SUMMARY:
Ziziphus honey can improve bone healing at extracted tooth sockets in humans by increasing salivary levels of bone markers, OPN and BMP-2.

DETAILED DESCRIPTION:
objectives of study: To study the effects of ziziphus honey on bone healing of extracted tooth socket in humans by comparing 1) Levels of BMP-2 and OPN in experimental and control groups at different intervals and 2) By radiographically measuring RBD of extraction sockets in experimental and control groups.

Aim of study: Post extraction ridge resorption is a major concern for future tooth prosthesis or implant placement. Honey can possibly help to improve bone healing and minimize ridge resorption after extractions.

Materials and Methods: Randomized controlled trial with simple random sampling of healthy individuals will be done. Total number of 30 participants will be equally divided into experimental group and control group. After tooth extractions in both groups, ziziphus honey will be injected into extracted sockets of experimental group while control group will be left as it is. Levels of BMP-2 and OPN will be tested in saliva through ELISA technique at day 0, 3 and 7 of tooth extraction and RBD will be measured on periapical radiographs at day 3, 21 and 40 in both groups.

Keywords: Bone morphogenetic protein-2 (BMP-2), Osteopontin (OPN), Relative bone density (RBD), Enzyme linked immunosorbent assay (ELISA).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy patients of either gender with adult age
2. No known hypersensitivity to honey.
3. Permanent maxillary or mandibular molars (first or second molars)

Exclusion Criteria:

1. History of radiotherapy or chemotherapy
2. Diabetic and hypertensive patients.
3. Pregnant and lactating females.
4. Smoking or consumption of alcohol
5. Bone conditions like osteoporosis etc.
6. Patients on oral contraceptives or steroid therapy
7. Subjects taking antibiotics or NSAIDS within one week.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
levels of BMP-2 | 1 week
  bone morphogenetic protein-2 levels to access amount of bone healing
levels of OPN | 1 week
  Osteopontin levels to access amount of bone healing
Relative bone density | 40 days
  bone quality confirmed on periapical radiographs in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Momina Khalid, BDS, Principal Investigator — PGMI, Lahore
Locations (1):
- Post graduate medical institute, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mendes RM, Silva GA, Lima MF, Calliari MV, Almeida AP, Alves JB, Ferreira AJ. Sodium hyaluronate accelerates the healing process in tooth sockets of rats. Arch Oral Biol. 2008 Dec;53(12):1155-62. doi: 10.1016/j.archoralbio.2008.07.001. Epub 2008 Aug 9. PMID 18692778
- See also: bone healing assessed through BMP-2 and OPN — https://pubmed.ncbi.nlm.nih.gov/18692778/